CLINICAL TRIAL: NCT05203341
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of NBI-1065845 in Adult Subjects With Major Depressive Disorder (MDD)
Brief Title: Study to Assess the Efficacy and Safety of NBI-1065845 in Adults With Major Depressive Disorder (MDD)
Acronym: SAVITRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-1065845-MDD2024; 2021-003989-12 (EudraCT Number)
Record Dates: First submitted 2021-11-18; First posted 2022-01-24 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Major Depressive Disorder
Keywords: Depression; MDD; Major Depressive Disorder; NBI-1065845; Mental Disorders; TAK-653; MADRS; SAVITRI
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive placebo orally once a day.
  Interventions: Drug: Placebo
- NBI-1065845 Low Dose (Experimental): Participants will receive low-dose NBI-1065845 orally once a day.
  Interventions: Drug: NBI-1065845
- NBI-1065845 High Dose (Experimental): Participants will receive high-dose NBI-1065845 orally once a day.
  Interventions: Drug: NBI-1065845

INTERVENTIONS:
Drug: Placebo — Matching placebo tablets
  Arms: Placebo
Drug: NBI-1065845 — NBI-1065845 tablets
  Other Names: TAK-653
  Arms: NBI-1065845 High Dose; NBI-1065845 Low Dose

SUMMARY:
The purpose of this study is to evaluate the efficacy of NBI-1065845 compared with placebo in participants with MDD on improving symptoms of depression.

ELIGIBILITY:
Key Inclusion Criteria:

Participants must meet all of these criteria for inclusion in the study:

1. The participant has completed written informed consent.
2. At the time of signing the informed consent, participant must be 18 to 65 years of age, inclusive.
3. The participant has a primary diagnosis of recurrent Major Depressive Disorder (MDD) or persistent depressive disorder.
4. Participant must have had inadequate response to antidepressant treatment.
5. Participant must have a Total Hamilton Depression Rating Scale-17 Item (HAMD-17) score ≥ 22 at screening.
6. Participants currently receiving pharmacological treatment for depression must have been taking current antidepressant medication(s) for ≥8 weeks prior to screening. Subjects not currently receiving pharmacologic treatment for depression must have received the most recent antidepressant medication(s) for ≥8 weeks in the current episode of depression.
7. Participants must be willing and able to comply with all study procedures.

Key Exclusion Criteria:

Participants will be excluded from the study if they meet any of the following criteria:

1. Participant is pregnant or breastfeeding or plans to become pregnant during the study.
2. Participant has an unstable medical condition or unstable chronic disease.
3. Participant has a history of neurological abnormalities.
4. Participant has a current or prior psychiatric disorder that was the primary focus of treatment other than MDD.
5. The participant's depressive symptoms have previously demonstrated nonresponse to an adequate course of treatment with electroconvulsive therapy (ECT).
6. The participant has an alcohol or substance use disorder.
7. In the Investigator's opinion, the participant is not capable of adhering to the protocol requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Total Montgomery Åsberg Depression Rating Scale (MADRS) Score at Day 28 | Baseline, Day 28

SECONDARY OUTCOMES:
Change from Baseline in Total MADRS Score at Day 7, Day 14, and Day 56 | Baseline, Days 7, 14, and 56
Change from Baseline in Clinical Global Impression - Severity (CGI-S) Score at Day 28 and Day 56 | Baseline, Days 28 and 56
Response, defined as ≥50% decrease in MADRS from baseline, at Day 28 and Day 56 | Baseline, Days 28 and 56
Remission, defined as MADRS ≤10, at Days 28 and 56 | Days 28 and 56
Change from Baseline in Patient Health Questionnaire-9 (PHQ-9) Score at Day 28 and Day 56 | Baseline, Days 28 and 56

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (39):
- United States (17):
  - Neurocrine Clinical Site, Birmingham, Alabama
  - Neurocrine Clinical Site, Huntsville, Alabama
  - Neurocrine Clinical Site, Riverside, California
  - Neurocrine Clinical Site, San Diego, California
  - Neurocrine Clinical Site, San Francisco, California
  - Neurocrine Clinical Site, Torrance, California
  - Neurocrine Clinical Site, Hartford, Connecticut
  - Neurocrine Clinical Site, Palmetto Bay, Florida
  - Neurocrine Clinical Site, Gaithersburg, Maryland
  - Neurocrine Clinical Site, Weldon Spring, Missouri
  - Neurocrine Clinical Site, Columbus, Ohio
  - Neurocrine Clinical Site, North Canton, Ohio
  - Neurocrine Clinical Site, Oklahoma City, Oklahoma
  - Neurocrine Clinical Site, Memphis, Tennessee
  - Neurocrine Clinical Site, Dallas, Texas
  - Neurocrine Clinical Site, Houston, Texas
  - Neurocrine Clinical Site, Draper, Utah
- Bulgaria (7):
  - Neurocrine Clinical Site, Plovdiv
  - Neurocrine Clinical Site, Rousse
  - Neurocrine Clinical Site, Sofia
  - Neurocrine Clinical Site, Tsarev Brod
  - Neurocrine Clinical Site, Varna
  - Neurocrine Clinical Site, Veliko Tarnovo
  - Neurocrine Clinical Site, Vratsa
- Czechia (3):
  - Neurocrine Clinical Site, Kladno
  - Neurocrine Clinical Site, Pilsen
  - Neurocrine Clinical Site, Prague
- Poland (4):
  - Neurocrine Clinical Site, Bełchatów
  - Neurocrine Clinical Site, Chełmno
  - Neurocrine Clinical Site, Gdansk
  - Neurocrine Clinical Site, Katowice
- Slovakia (4):
  - Neurocrine Clinical Site, Košice
  - Neurocrine Clinical Site, Rimavská Sobota
  - Neurocrine Clinical Site, Trenčín
  - Neurocrine Clinical Site, Vranov nad Topľou
- Sweden (4):
  - Neurocrine Clinical Site, Gothenburg
  - Neurocrine Clinical Site, Halmstad
  - Neurocrine Clinical Site, Lund
  - Neurocrine Clinical Site, Stockholm

IPD SHARING:
Plan to Share IPD: No